CLINICAL TRIAL: NCT02936323
Title: A Phase 1/2a, Open-label Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of PEN-221 in Patients With Somatostatin Receptor 2 Expressing Advanced Cancers, Including Gastroenteropancreatic or Lung or Thymus or Other Neuroendocrine Tumors or Small Cell Lung Cancer or Large Cell Neuroendocrine Carcinoma of the Lung
Brief Title: PEN-221 in Somatostatin Receptor 2 Expressing Advanced Cancers Including Neuroendocrine and Small Cell Lung Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tarveda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PEN-221-001
Record Dates: First submitted 2016-10-13; First posted 2016-10-18 (Estimated); Results first posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Neuroendocrine Tumors; Carcinoma, Small Cell Lung; Neuroendocrine Carcinoma
Keywords: SCLC small cell lung cancer; pancreatic neuroendocrine NET; GI neuroendocrine NET
MeSH Terms: conditions — Neuroendocrine Tumors; Small Cell Lung Carcinoma; Carcinoma, Neuroendocrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1: Dose Escalation (Experimental): Cohort 1 will consist of two (2) participants who will receive PEN-221 at the starting dose of 1.0 mg. The first participant will be followed for at least 7 days for safety and dose limiting toxicity (DLT). If PEN-221 is tolerated, the second participant will be enrolled into the cohort. The two (2) participants will be followed for safety and DLTs for at least a 4-week observation period. The Safety Review Committee (SRC) will determine the initiation of cohort 2.
  Cohort 2 and each subsequent dose escalation cohort will consist of 3 to 6 participants who will be treated at each dose level of PEN-221 as determined by the SRC and will be followed for safety and DLTs for at least a 3-week observation period. Each dose escalation level and cohort initiation will be determined by the SRC.
  Dose escalation will continue until the Maximum Tolerated Dose (MTD) of PEN-221 is determined and the Recommended Phase 2a Dose (RP2D) is established by the SRC.
  Interventions: Drug: PEN-221
- Phase 2a: Dose Expansion (GI mid-gut NET) (Experimental): Gastrointestinal mid-gut NET Cohort
  Interventions: Drug: PEN-221
- Phase 2a: Dose Expansion (PNET) (Experimental): Pancreatic NET Cohort
  Interventions: Drug: PEN-221
- Phase 2a: Dose Expansion (SCLC) (Experimental): Small Cell Lung Cancer Cohort
  Interventions: Drug: PEN-221

INTERVENTIONS:
Drug: PEN-221 — PEN-221 administered IV over 1 hour on an every 3-week cycle (21 days +/- 2 days) starting dose of 1 mg with each subsequent cohort increased starting dose level until MTD is reached.
  Arms: Phase 1: Dose Escalation
Drug: PEN-221 — PEN-221 administered IV over 1 hour on an every 3-week cycle (21 days +/- 2 days) starting dose at recommended Phase 2a dose established in Phase 1.
  Arms: Phase 2a: Dose Expansion (GI mid-gut NET); Phase 2a: Dose Expansion (PNET); Phase 2a: Dose Expansion (SCLC)

SUMMARY:
Protocol PEN-221-001 is an open-label, multicenter Phase 1/2a study evaluating PEN-221 in patients with SSTR2 expressing advanced gastroenteropancreatic (GEP) or lung or thymus or other neuroendocrine tumors or small cell lung cancer or large cell neuroendocrine carcinoma of the lung.

DETAILED DESCRIPTION:
Protocol PEN-221-001 will first enroll patients into a dose escalation phase, where a Bayesian logistic regression model, guided by the escalation with overdose control principle and overseen by a safety review committee, will be used to make dose recommendations and estimate the maximum tolerated dose (MTD).

Once the MTD has been confirmed, remaining patients will be enrolled into a full expansion phase to assess PEN-221 efficacy in patients with gastrointestinal mid-gut neuroendocrine tumors or pancreatic neuroendocrine tumors or small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* M/F at least 18 years old
* ECOG performance status 0 or 1
* Adequate bone marrow, liver, and kidney function within 2 weeks prior to first dose
* Serum potassium, calcium, magnesium, phosphorus within normal limits (may be supplemented)
* Adequate birth control
* Somatostatin receptor 2 positive tumor as assessed at pre-screening or within 180 d of first drug dose using indium SPECT or gallium PET

Patients in Phase 1 must have a histologically or cytologically-confirmed solid tumor in 1 of the following categories:

* Advanced small cell lung cancer (SCLC) or large cell neuroendocrine carcinoma (LCNEC) of lung progressed after at least 1 line of anticancer chemotherapy
* Advanced low or intermediate grade gastroenteropancreatic or lung or thymus neuroendocrine tumor (NET), or NET of unknown primary, progressed after at least 1 line of anticancer therapy (unless no standard treatments available or such treatments are deemed not appropriate)
* Advanced paraganglioma, pheochromocytoma, medullary thyroid carcinoma, Merkel cell carcinoma, or high grade extrapulmonary neuroendocrine carcinoma having progressed after 1 or more lines of anticancer chemotherapy (unless no standard treatments available or such treatments are deemed not appropriate)

For patients enrolling once escalation is complete (Phase 2a), disease must be measurable per RECIST 1.1 criteria with last imaging performed within 28 days prior to first drug dose

In addition to the criterion listed above, Patients in Phase 2a must have a histologically- or cytologically-confirmed, advanced or metastatic solid tumor, in 1 of the following categories: disease history specified in one of the criteria listed below:

* Well differentiated, low or intermediate grade, gastrointestinal mid-gut (arising from the lower jejunum, ileum, appendix, cecum, and proximal colon) NET with documented disease progression within 6 months prior to start of study treatment and evidence of radiographic disease progression based on scans performed not more than 15 months apart. Patients may have received 1 or more prior lines of anticancer therapy, such as somatostatin analogues, targeted agents, or liver-directed intra-arterial therapy, but are NOT eligible if they have received prior systemic cytotoxic chemotherapy.
* Well differentiated, low or intermediate grade, pancreatic NET with documented disease progression within 6 months prior to start of study treatment and evidence of radiographic disease progression based on scans performed not more than 15 months apart. Patients may have received 1 or more prior lines of anticancer therapy, such as somatostatin analogues, targeted agents, or liver-directed intra-arterial therapy, and up to 1 prior line of systemic cytotoxic chemotherapy, but are NOT eligible if they have received more than 1 prior line of systemic cytotoxic chemotherapy or if they have received prior peptide receptor radionuclide therapy (PRRT)
* SCLC after having received up to three prior lines of anticancer therapy.

Exclusion Criteria:

* Treatment with anticancer therapy or investigational drug or device within 3 wk (6 wk for nitrosureas or mitomycin C) or 5 half-lives of agent, whichever is shorter, prior to first PEN-221 drug dose, and any drug-related toxicities must have recovered to grade 1 or less
* Any other malignancy known to be active or treated within 3 years of start of screening, except cervical intra-epithelial neoplasia, superficial (non-invasive) bladder cancer, and non-melanoma skin cancer
* Cardiac criteria such as unstable angina, myocardial infarction within 6 months of screening, NY Heart Association Class 1 or 2 heart failure, QTc greater than 470 msec, congenital long Qt syndrome, symptomatic orthostatic hypotension within 6 months of screening, uncontrolled hypertension, or clinically important abnormalities in heart rhythm, conduction, morphology of resting ECG
* Stroke or transient ischemic attack within 6 months of screening
* Peripheral neuropathy greater than grade 1
* Requirement for medication with strong CYP3A4 inhibitor
* History of leptomeningeal disease or spinal cord compression
* Brain metastases unless asymptomatic on a stable low dose of steroids. Patients with SCLC or LCNEC of lung only must have CT or MRI of brain during screening, and if metastases found, must have radiotherapy with 14 day washout or stereotactic radiotherapy or radio surgery with 7 day washout prior to first drug dose.
* Major surgery within 28 days of first drug dose
* Female who is pregnant or breast feeding
* Evidence of severe uncontrolled systemic disease, bleeding diatheses, renal or liver transplant, active infection with hepatitis B or C, or HIV
* Hypersensitivity or anaphylactic reaction to any somatostatin analog or to maytansinoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Tarveda Therapeutics
Locations (13):
- United States (10):
  - Florida Cancer Specialists South, Fort Myers, Florida
  - Florida Cancer Specialists North, St. Petersburg, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center/ NY Presbyterian, Manhattan, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Sarah Cannon Research Institute/Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- United Kingdom (3):
  - University College London, London
  - The Christie NHS Trust, Manchester
  - Southampton General Hospital, Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled with SSTR2 expressing advanced gastroenteropancreatic or lung or thymus or other NETs or SCLC or LCNEC of the lung. A total of 23 participants enrolled into the Phase 1 Dose Escalation stage of the study receiving at least one dose of PEN-221 and a total of 66 patients enrolled into the Phase 2a Disease-Specific Dose Expansion stage of the study receiving at least one dose of PEN-221.
Pre-assignment Details: Each eligible participant must have demonstrated a tumor that was positive for expression of SSTR2 by historical or study-related somatostatin analog radioimaging (SARI). Participants who discontinued treatment entered a follow-up period (Disease Progression Follow-up and/or Long-Term Follow-up). Results for data collected up to cut-off 31 July 2020 are reported here.
Groups:
- Phase 1 Dose Escalation (Cohort 1): Participants in Cohort 1 received PEN-221 administered IV over 1 hour at the starting dose of 1.0 mg on an every 3-week cycle (21 days +/-2 days).
- Phase 1 Dose Escalation (Cohort 2): Participants in Cohort 2 received PEN-221 administered IV over 1 hour at the starting dose of 2.0 mg on an every 3-week cycle (21 days +/-2 days).
- Phase 1 Dose Escalation (Cohort 3): Participants in Cohort 3 received PEN-221 administered IV over 1 hour at the starting dose of 4.0 mg on an every 3-week cycle (21 days +/-2 days).
- Phase 1 Dose Escalation (Cohort 4): Participants in Cohort 4 received PEN-221 administered IV over 1 hour at the starting dose of 8.0 mg on an every 3-week cycle (21 days +/-2 days).
- Phase 1 Dose Escalation (Cohort 5): Participants in Cohort 5 received PEN-221 administered IV over 1 hour at the starting dose of 12.0 mg on an every 3-week cycle (21 days +/-2 days).
- Phase 1 Dose Escalation (Cohort 6): Participants in Cohort 6 received PEN-221 administered IV over 1 hour at the starting dose of 18.0 mg on an every 3-week cycle (21 days +/-2 days).
- Phase 1 Dose Escalation (Cohort 7): Participants in Cohort 7 received PEN-221 administered IV over 1 hour at the starting dose of 25.0 mg on an every 3-week cycle (21 days +/-2 days).
- Phase 2a Dose Expansion (GI Mid-gut NET Cohort): Participants were enrolled with advanced or metastatic, well-differentiated, low or intermediate grade gastrointestinal mid-gut Neuroendocrine Tumor (GINET).
  Participants in the GINET cohort were enrolled into one of two groups which included 25 participants without prior Peptide Receptor Radionuclide Therapy [PRRT] (GINET PRRT Naïve) and 7 participants with prior PRRT (GINET PRRT Recurrent).
- Phase 2a Dose Expansion (PNET Cohort): Participants were enrolled with advanced or metastatic, well-differentiated, low or intermediate grade pancreatic Neuroendocrine Tumor (PNET).
- Phase 2a Dose Expansion (SCLC Cohort): Participants were enrolled with advanced or metastatic Small Cell Lung Cancer (SCLC).
Period: Phase 1 Dose Escalation
Arm/Group | Phase 1 Dose Escalation (Cohort 1) | Phase 1 Dose Escalation (Cohort 2) | Phase 1 Dose Escalation (Cohort 3) | Phase 1 Dose Escalation (Cohort 4) | Phase 1 Dose Escalation (Cohort 5) | Phase 1 Dose Escalation (Cohort 6) | Phase 1 Dose Escalation (Cohort 7) | Phase 2a Dose Expansion (GI Mid-gut NET Cohort) | Phase 2a Dose Expansion (PNET Cohort) | Phase 2a Dose Expansion (SCLC Cohort)
Started | 2 (Participants in Phase 1 did not advance to Phase 2a.) | 3 (Participants in Phase 1 did not advance to Phase 2a.) | 3 (Participants in Phase 1 did not advance to Phase 2a.) | 3 (Participants in Phase 1 did not advance to Phase 2a.) | 3 (Participants in Phase 1 did not advance to Phase 2a.) | 6 (Participants in Phase 1 did not advance to Phase 2a.) | 3 (Participants in Phase 1 did not advance to Phase 2a.) | 0 | 0 | 0
Completed (Participants in the follow-up period of Phase 1 study as of data cut-off date 31 Jul 2020.) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not Completed | 2 | 2 | 3 | 2 | 3 | 5 | 3 | 0 | 0 | 0
Not completed — Informed Consent Withdrawn | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 1 | 3 | 1 | 2 | 3 | 3 | 0 | 0 | 0
Not completed — Study Discontinued at Site | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Phase 2a Dose Expansion
Arm/Group | Phase 1 Dose Escalation (Cohort 1) | Phase 1 Dose Escalation (Cohort 2) | Phase 1 Dose Escalation (Cohort 3) | Phase 1 Dose Escalation (Cohort 4) | Phase 1 Dose Escalation (Cohort 5) | Phase 1 Dose Escalation (Cohort 6) | Phase 1 Dose Escalation (Cohort 7) | Phase 2a Dose Expansion (GI Mid-gut NET Cohort) | Phase 2a Dose Expansion (PNET Cohort) | Phase 2a Dose Expansion (SCLC Cohort)
Started (Initial Phase 2a PEN-221 start dose at Phase 1 MTD and RP2D of 18 mg flat dose. After review of 19 Phase 2a participants, SRC decreased start dose from 18 mg to 15 mg flat dose due to higher-than-expected treatment discontinuation rate. After review of all Phase 1 and 31 Phase 2a participants, SRC changed 15 mg flat dose to Body Surface Area (BSA) based PEN-221 dose of 8.8 mg/m^2 due to correlation between BSA and drug exposure (AUC) associated with higher rate of participant discontinuation.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 32 (Participants in Phase 2a did not participate in Phase 1) | 15 (Participants in Phase 2a did not participate in Phase 1) | 19 (Participants in Phase 2a did not participate in Phase 1)
Completed (Participants in the follow-up period of Phase 2a study as of data cut-off date 31 Jul 2020.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 2 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 13 | 14
Not completed — Informed Consent Withdrawn | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 4 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Change(s) to patient's condition | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 10

BASELINE CHARACTERISTICS:
Population: The analysis population was the Full Analysis Set (FAS) which consisted of all participants enrolled into the study and who receive any amount of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Escalation (Cohort 1) | Phase 1 Dose Escalation (Cohort 2) | Phase 1 Dose Escalation (Cohort 3) | Phase 1 Dose Escalation (Cohort 4) | Phase 1 Dose Escalation (Cohort 5) | Phase 1 Dose Escalation (Cohort 6) | Phase 1 Dose Escalation (Cohort 7) | Phase 2a Dose Expansion (GI Mid-gut NET Cohort) | Phase 2a Dose Expansion (PNET Cohort) | Phase 2a Dose Expansion (SCLC Cohort) | Total
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 6 | 3 | 32 | 15 | 19 | 89
Age, Continuous [Median (Full Range); unit: Years] | 48.5 [40 to 57] | 57.0 [54 to 74] | 67.0 [43 to 69] | 46.0 [33 to 71] | 67.0 [57 to 69] | 63.5 [45 to 67] | 52.0 [27 to 73] | 66.0 [32 to 81] | 58.0 [36 to 77] | 65.0 [39 to 82] | 65 [27 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 1 | 2 | 3 | 2 | 15 | 8 | 10 | 43
  Male | 2 | 3 | 1 | 2 | 1 | 3 | 1 | 17 | 7 | 9 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 2 | 2 | 3 | 3 | 1 | 6 | 3 | 27 | 10 | 19 | 76
  Black | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 6
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Native American or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not collected | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 6
  Not Hispanic or Latino | 1 | 3 | 3 | 3 | 2 | 5 | 2 | 30 | 13 | 19 | 81
  Not collected | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose of PEN-221 and Recommended Phase 2a Dose (RP2D)
Description: MTD was determined by testing increasing doses up to 25 mg flat dose IV over 1 hour on an every 3 week cycle on dose escalation cohorts 1 to 7 with 2 participants in cohort 1 and 3-6 participants each in cohorts 2-7. The MTD was defined as the highest drug dosage not causing a Dose Limiting Toxicity (DLT) in > 33% of the treated participants during the first cycle of treatment. DLTs were defined as any Grade 3 or 4 adverse event (AE) using the Common Terminology Criteria for Adverse Events Version 4.03 occurring within the first 4 weeks for cohort 1 and within 3 weeks for each subsequent cohort that was not related to underlying disease, disease progression, intercurrent illness, or concomitant medications. The RP2D was established by achieving the Maximum Tolerated Dose (MTD). The RP2D may be equal to or below the MTD.
Time Frame: Up to 4 weeks in the first cohort and up to 3 weeks for each subsequent cohort
Population: All Phase 1 participants who received at least one dose of PEN-221 and either experienced a DLT or had been followed for the full DLT evaluation period.
Measure: Number; unit: mg
Groups:
- All Participants in Phase 1 Dose Escalation (Cohorts 1-7): All participants who received at least 1 dose of PEN-221, either at 1.0 mg, 2.0 mg, 4.0 mg, 8.0 mg, 12.0 mg, 18.0 mg, 25.0 mg via IV.
Arm/Group | All Participants in Phase 1 Dose Escalation (Cohorts 1-7)
Number analyzed (Participants) | 23
mg | 18.0

2. Primary Outcome: Phase 1: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: DLTs were defined as any Grade 3 or 4 adverse event (AE) using the Common Terminology Criteria for Adverse Events Version 4.03 occurring within the first 4 weeks for cohort 1 and within 3 weeks for each subsequent cohort that was not related to underlying disease, disease progression, intercurrent illness, or concomitant medications. Grade 3 is a severe AE and Grade 4 is a life-threatening or disabling AE. DLTs were collected to determine the Maximum-Tolerated Dose (MTD), which is defined as the dose level below the dose at which > 33% of participants experienced a DLT during the first cycle of treatment.
Time Frame: Up to 4 weeks in the first cohort and up to 3 weeks for each subsequent cohort
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Phase 1 Dose Escalation (Cohort 1) | Phase 1 Dose Escalation (Cohort 2) | Phase 1 Dose Escalation (Cohort 3) | Phase 1 Dose Escalation (Cohort 4) | Phase 1 Dose Escalation (Cohort 5) | Phase 1 Dose Escalation (Cohort 6) | Phase 1 Dose Escalation (Cohort 7)
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 6 | 3
participants | 0 | 0 | 0 | 0 | 0 | 0 | 2

3. Primary Outcome: Phase 2a: Percentage of Gastrointestinal Mid-gut NETs and Pancreatic NETs Participants Who Achieved Clinical Benefit as Determined by RECIST 1.1
Description: Efficacy of PEN-221 in gastrointestinal mid-gut NETs and pancreatic NETs using clinical benefit rate (CBR) defined as the best overall response of complete response (CR), partial response (PR), or stable disease (SD) according to RECIST 1.1 using the investigator assessment.
Time Frame: Baseline and every 9 weeks up to time of disease progression (per RECIST 1.1) or death, up to data cut-off (31 Jul 2020).
Population: Outcome measured by cancer type. GI mid-gut NET or PNET participants who received any amount of study drug and had at least 1 post-baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 2a Dose Expansion (PNET Cohort: Participants were enrolled with advanced or metastatic, well-differentiated, low or intermediate grade pancreatic Neuroendocrine Tumor (PNET).
Arm/Group | Phase 2a Dose Expansion (GI Mid-gut NET Cohort) | Phase 2a Dose Expansion (PNET Cohort
Number analyzed (Participants) | 26 | 12
percentage of participants | 88.5 [69.8 to 97.6] | 50 [21.1 to 78.9]

4. Primary Outcome: Phase 2a: Number of Small Cell Lung Cancer (SCLC) Participants Who Achieved an Objective Response of Complete Response (CR) or Partial Response (PR) as Defined by RECIST 1.1.
Description: Efficacy of PEN-221 in Small Cell Lung Cancer (SCLC) using objective response rate (ORR) as defined as the best overall response of CR or PR using tumor response criteria defined by RECIST 1.1.
Time Frame: Baseline and every 6 weeks up to time of disease progression (per RECIST 1.1) or death, up to data cut-off (31 Jul 2020).
Population: Outcome measured by cancer type. SCLC participants who received any amount of study drug and had at least 1 post-baseline efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2a Dose Expansion (SCLC Cohort)
Number analyzed (Participants) | 12
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 3
  Progressive Disease | 9

5. Primary Outcome: Phase 2a: Duration of Response (DOR) for Small Cell Lung Cancer (SCLC)
Description: Duration of Response (DOR) is defined as the time from the first documented response (CR or PR), as assessed by the investigator, to the date of first documented disease progression or death due to underlying cancer. If patient did not progress or die before the data cutoff date (31-July-2020), DOR was censored at the date of last adequate tumor assessment.
Time Frame: From the date of first treatment through the date of first documented progression, assessed up to data cut-off (31 Jul 2020).
Population: Outcome measured by cancer type. SCLC participants who received any amount of study drug and had at least 1 post-baseline efficacy assessment. No participants in the SCLC cohort had an objective response, so no data is presented for this Outcome Measure.
Groups:
- Phase 2a Dose Expansion (SCLC Cohort): Outcome measured by cancer type. SCLC participants who received any amount of study drug and had at least 1 post-baseline efficacy assessment. No participants in the SCLC cohort had an objective response, so no data is presented for this Outcome Measure.
Arm/Group | Phase 2a Dose Expansion (SCLC Cohort)
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Study Participants Who Experienced Treatment-Emergent Adverse Events
Description: Phase 1 and Phase 2a participants who experienced any Treatment-Emergent Adverse Event (TEAE) to determine the safety and tolerability of PEN-221. TEAEs are any AE that occurred after first dose of study drug through 28 days after the last dose of study drug, any event considered study drug related regardless of start date of the event, or any event that was present at baseline but worsened in intensity or was subsequently considered study drug related by the Investigator. Phase 2a TEAEs were collected for reporting in the BSA dosing format only.
Time Frame: From date of first treatment/trial entry until 28 days after last treatment for each participant, up to data cut-off (31 Jul 2020).
Population: The Safety Analysis population was comprised of all enrolled participants who received any amount of study drug and had at least 1 post-baseline safety evaluation. All non-BSA based doses in Phase 2a were converted to BSA dosing units.
  Participants dosed under the initial MTD dosing regimen were assigned to the < 8.8 mg/m^2 or > 8.8 mg/m^2 dose groups based on the BSA conversion of the initial study dose.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2a Dose Expansion (<8.8 mg/m^2): Participants in GINET, PNET, and SCLC received PEN-221 BSA calculated starting dose of less than 8.8 mg/m^2 on an every 3-week cycle (21 days +/-2 days)
  All non-BSA based doses in Phase 2a were converted to BSA dosing units. Participants dosed under the initial MTD dosing regimen were assigned to the < 8.8 mg/m^2 or > 8.8 mg/m^2 dose groups based on the BSA conversion of the initial study dose.
- Phase 2a Dose Expansion (8.8 mg/m^2): Participants in GINET, PNET, and SCLC received PEN-221 BSA starting dose of 8.8 mg/m^2 on an every 3-week cycle (21 days +/-2 days)
- Phase 2a Dose Expansion (>8.8 mg/m^2): Participants in GINET, PNET, and SCLC received PEN-221 BSA calculated starting dose of more than 8.8 mg/m^2 on an every 3-week cycle (21 days +/-2 days)
  All non-BSA based doses in Phase 2a were converted to BSA dosing units. Participants dosed under the initial MTD dosing regimen were assigned to the < 8.8 mg/m^2 or > 8.8 mg/m^2 dose groups based on the BSA conversion of the initial study dose.
Arm/Group | Phase 1 Dose Escalation (Cohort 1) | Phase 1 Dose Escalation (Cohort 2) | Phase 1 Dose Escalation (Cohort 3) | Phase 1 Dose Escalation (Cohort 4) | Phase 1 Dose Escalation (Cohort 5) | Phase 1 Dose Escalation (Cohort 6) | Phase 1 Dose Escalation (Cohort 7) | Phase 2a Dose Expansion (<8.8 mg/m^2) | Phase 2a Dose Expansion (8.8 mg/m^2) | Phase 2a Dose Expansion (>8.8 mg/m^2)
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 6 | 3 | 12 | 34 | 20
Participants
  Any TEAE | 2 | 3 | 3 | 3 | 3 | 6 | 3 | 12 | 32 | 20
  Serious TEAEs | 2 | 1 | 3 | 0 | 0 | 2 | 2 | 3 | 7 | 15
  Treatment Related TEAEs | 0 | 3 | 3 | 3 | 3 | 6 | 3 | 10 | 29 | 19
  TEAEs leading to Discontinuation of Study Drug | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 7 | 6
  TEAEs leading to Death | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Dose Limiting Toxicity | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0

7. Secondary Outcome: Maximum Concentration (Cmax) of PEN-221, DM1, and Peptide
Description: Blood samples were obtained and plasma concentrations were determined using validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) methods. Phase 2a data were collected for reporting in the BSA dosing format only.
Time Frame: Phase 1: Day 1 of Cycles 1 and 3 pre-start of infusion (SOI), at 0.5, 1, 1.5, 2, 4, 6, 8, 10 hours post-start of infusion. Phase 2a: Day 1 Cycle 1 pre-start of infusion, at 0.5,1, 1.5, 2, 4, 6, 8, 24 hours post-SOI; once at Day 8 Cycle 1.
Population: The Pharmacokinetic Analysis set comprises all participants who received any amount of study drug and provided adequate PK samples.
  Phase 2a participants dosed under the initial MTD dosing regimen were assigned to the < 8.8 mg/m^2 or > 8.8 mg/m^2 dose groups based on the BSA conversion of the initial study dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1 Dose Escalation (Cohort 1) | Phase 1 Dose Escalation (Cohort 2) | Phase 1 Dose Escalation (Cohort 3) | Phase 1 Dose Escalation (Cohort 4) | Phase 1 Dose Escalation (Cohort 5) | Phase 1 Dose Escalation (Cohort 6) | Phase 1 Dose Escalation (Cohort 7) | Phase 2a Dose Expansion (<8.8 mg/m^2) | Phase 2a Dose Expansion (8.8 mg/m^2) | Phase 2a Dose Expansion (>8.8 mg/m^2)
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 6 | 3 | 12 | 28 | 20
ng/mL
  Plasma PK | 18.96 (9.56) | 50.20 (24.30) | 150.40 (51.99) | 359.70 (92.42) | 592.50 (149.66) | 2802 (5068.6) | 1324 (519.94) | 451.4 (174.14) | 1533 (3356.9) | 1064 (2298.7)
  Total Peptide | 16.38 (3.7112) | 40.03 (15.807) | 129.8 (5.7813) | 261.4 (49.269) | 420.2 (69.703) | 1925 (3246.8) | 926.9 (279.02) | 350.0 (102.28) | 1041 (2061.0) | 831.5 (1721.0)
  Total DM1 | 11.11 (2.7669) | 29.88 (14.304) | 94.01 (2.7951) | 198.6 (37.848) | 340.4 (87.602) | 1327 (2157.2) | 691.3 (165.22) | 261.2 (70.449) | 762.3 (1388.0) | 505.9 (734.05)
  Unconjugated DM1 | 4.758 (0.78830) | 13.79 (6.1768) | 42.23 (12.295) | 78.63 (6.2100) | 112.0 (22.186) | 218.3 (73.574) | 266.3 (46.561) | 101.0 (26.560) | 164.5 (74.435) | 146.3 (74.755)
  Free Sulfhydryl DM1: number analyzed (Participants) | 2 | 3 | 2 | 2 | 3 | 6 | 3 | 10 | 28 | 19
  Free Sulfhydryl DM1 | 0.09568 (0.034873) | 0.2441 (0.17198) | 0.6778 (0.02297) | 1.975 (0.46462) | 2.739 (0.90804) | 14.12 (18.151) | 11.04 (5.011) | 2.174 (0.82698) | 5.214 (8.2827) | 6.225 (12.276)

8. Secondary Outcome: Area Under the Curve (AUC) of PEN-221, DM1, and Peptide
Description: as for outcome 7
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: (ng/mL)*h
Arm/Group | Phase 1 Dose Escalation (Cohort 1) | Phase 1 Dose Escalation (Cohort 2) | Phase 1 Dose Escalation (Cohort 3) | Phase 1 Dose Escalation (Cohort 4) | Phase 1 Dose Escalation (Cohort 5) | Phase 1 Dose Escalation (Cohort 6) | Phase 1 Dose Escalation (Cohort 7) | Phase 2a Dose Expansion (<8.8 mg/m^2) | Phase 2a Dose Expansion (8.8 mg/m^2) | Phase 2a Dose Expansion (>8.8 mg/m^2)
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 6 | 3 | 12 | 28 | 20
(ng/mL)*h
  Plasma PK: number analyzed (Participants) | 2 | 3 | 2 | 3 | 3 | 5 | 3 | 12 | 25 | 17
  Plasma PK | 38.34 (15.88) | 89.95 (33.64) | 192.40 (48.66) | 643.60 (224.39) | 1119 (330.86) | 2323 (2267.7) | 2357 (798.60) | 867.7 (329.9) | 1667 (1638.6) | 1463 (1141.8)
  Total Peptide: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 6 | 2 | 12 | 26 | 19
  Total Peptide | 87.20 (30.636) | 189.2 (64.194) | 548.0 (156.34) | 1080 (197.69) | 1730 (475.69) | 3147 (1211.0) | 4402 (938.17) | 2988 (847.68) | 4203 (1837.2) | 4558 (1474.5)
  Total DM1: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 4 | 2 | 11 | 24 | 16
  Total DM1 | 65.59 (16.501) | 179.7 (97.376) | 454.8 (136.89) | 981.1 (74.477) | 1780 (652.3) | 1996 (489.18) | 3980 (1335.4) | 2153 (526.06) | 3328 (1881.7) | 3419 (1277.9)
  Unconjugated DM1: number analyzed (Participants) | 2 | 3 | 2 | 2 | 1 | 4 | 1 | 11 | 20 | 15
  Unconjugated DM1 | 54.18 (15.810) | 163.9 (86.594) | 444.5 (100.94) | 720.6 (86.063) | 1384 | 1776 (660.31) | 4316 | 1765 (415.63) | 2384 (522.17) | 2781 (1057.1)
  Free Sulfhydryl DM1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 4 | 3 | 8 | 21 | 15
  Free Sulfhydryl DM1 |  |  |  | 16.86 | 17.63 (7.6946) | 37.40 (12.335) | 131.4 (109.56) | 32.06 (20.012) | 62.05 (35.792) | 69.48 (58.396)

9. Secondary Outcome: Half-life (t1/2) of PEN-221, DM1, and Peptide
Description: Blood samples were obtained and plasma concentrations were determined using validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) methods. Phase 2a data collected for reporting in the BSA dosing format only.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1 Dose Escalation (Cohort 1) | Phase 1 Dose Escalation (Cohort 2) | Phase 1 Dose Escalation (Cohort 3) | Phase 1 Dose Escalation (Cohort 4) | Phase 1 Dose Escalation (Cohort 5) | Phase 1 Dose Escalation (Cohort 6) | Phase 1 Dose Escalation (Cohort 7) | Phase 2a Dose Expansion (<8.8 mg/m^2) | Phase 2a Dose Expansion (8.8 mg/m^2) | Phase 2a Dose Expansion (>8.8 mg/m^2)
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 6 | 3 | 12 | 28 | 20
hours
  Plasma PK: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 3 | 12 | 25 | 17
  Plasma PK | 1.46 [1.15 to 1.77] | 1.41 [1.31 to 1.80] | 1.77 [0.86 to 2.69] | 1.70 [1.59 to 2.32] | 1.94 [1.80 to 3.76] | 1.61 [1.26 to 3.64] | 3.06 [2.50 to 3.45] | 4.259 [1.04 to 9.01] | 4.180 [1.64 to 12.9] | 4.526 [1.27 to 6.93]
  Total Peptide: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 6 | 2 | 12 | 26 | 19
  Total Peptide | 5.33 [3.87 to 6.80] | 4.61 [4.15 to 5.29] | 5.25 [2.56 to 6.50] | 4.33 [3.61 to 5.57] | 5.63 [3.03 to 8.07] | 4.89 [2.27 to 11.2] | 7.49 [7.32 to 7.67] | 27.9 [10.1 to 35.0] | 28.7 [6.71 to 35.8] | 30.9 [22.9 to 38.6]
  Total DM1: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 4 | 2 | 11 | 24 | 16
  Total DM1 | 4.78 [3.61 to 5.94] | 4.48 [3.85 to 7.35] | 5.87 [2.94 to 6.13] | 4.43 [4.19 to 4.49] | 5.69 [3.25 to 9.13] | 5.43 [3.67 to 6.38] | 6.32 [5.66 to 6.98] | 25.3 [7.26 to 28.4] | 24.2 [5.57 to 27.6] | 25.5 [19.9 to 34.1]
  Unconjugated DM1: number analyzed (Participants) | 2 | 3 | 2 | 2 | 1 | 4 | 1 | 11 | 20 | 15
  Unconjugated DM1 | 5.77 [3.61 to 7.92] | 7.80 [6.38 to 9.00] | 6.07 [5.58 to 6.56] | 5.36 [4.73 to 5.98] | 8.49 [8.49 to 8.49] | 6.89 [4.67 to 9.60] | 8.94 [8.94 to 8.94] | 25.9 [6.98 to 29.4] | 24.5 [8.03 to 29.2] | 25.0 [19.8 to 34.8]
  Free Sulfhydryl DM1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 4 | 3 | 8 | 21 | 15
  Free Sulfhydryl DM1 |  |  |  | 4.57 | 4.93 [4.40 to 5.47] | 3.87 [2.57 to 4.21] | 9.01 [7.10 to 10.8] | 10.1 [6.22 to 38.1] | 20.9 [7.21 to 46.9] | 14.3 [8.16 to 47.2]

10. Secondary Outcome: Phase 1: Number of Participants With a Best Response of an Objective Response, Stable Disease, or Progressive Disease.
Description: Assess the potential of preliminary anti-tumor activity of PEN-221 using tumor response criteria as defined by RECIST 1.1.
Time Frame: Baseline, every 6 or 9 weeks depending on the tumor type, up to time of disease progression (per RECIST 1.1) or death, up to data cut-off (31 Jul 2020).
Population: Phase 1 participants who received at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation (Cohort 1) | Phase 1 Dose Escalation (Cohort 2) | Phase 1 Dose Escalation (Cohort 3) | Phase 1 Dose Escalation (Cohort 4) | Phase 1 Dose Escalation (Cohort 5) | Phase 1 Dose Escalation (Cohort 6) | Phase 1 Dose Escalation (Cohort 7)
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 3 | 6 | 2
Participants
  Complete Response (Confirmed or Unconfirmed) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (Confirmed) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (Unconfirmed) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Stable Disease | 1 | 3 | 1 | 3 | 2 | 2 | 2
  Progressive Disease | 1 | 0 | 0 | 0 | 1 | 4 | 0

11. Secondary Outcome: Phase 2a: Maximum Tolerated Dose (MTD) and Recommended Phase 2a Dose (RP2D) Based on Body Surface Area
Description: Confirm the MTD identified during the dose-escalation phase and further investigate the safety and tolerability of the RP2D and schedule of PEN-221. Initial Phase 2a PEN-221 start dose at Phase 1 MTD and RP2D was determined at 18 mg flat dose. The MTD was defined as the highest drug dosage not causing a Dose Limiting Toxicity (DLT) in > 33% of the treated participants during the first cycle of treatment. DLTs were defined as any Grade 3 or 4 adverse event (AE) using the Common Terminology Criteria for Adverse Events Version 4.03 occurring within the first 4 weeks for cohort 1 and within 3 weeks for each subsequent cohort that was not related to underlying disease, disease progression, intercurrent illness, or concomitant medications. The RP2D was established by achieving the Maximum Tolerated Dose (MTD). The RP2D may be equal to or below the MTD.
Time Frame: From date of first treatment/trial entry until 28 days after last treatment for each Phase 2a participant, up to data cut-off (31 Jul 2020)
Population: All Phase 2a participants who received any amount of study drug and had at least 1 post-baseline safety evaluation. SRC reviewed all Phase 1 and 31 Phase 2a participants and changed flat dose (mg) to Body Surface Area (BSA) based dose of 8.8 mg/m^2 due to correlation between BSA and drug exposure associated with higher rate of participant discontinuation. Calculated BSA capped at 2.0 m^2 so not to exceed Phase 1 MTD of 18 mg. Phase 2a data collected for reporting in the BSA dosing format only.
Measure: Number; unit: mg/m^2
Groups:
- All Phase 2a Dose Expansion Participants: All GINET, PNET, and SCLC participants who received at least 1 PEN-221 BSA calculated starting dose of either < 8.8 mg/m^2, 8.8 mg/m^2, or > 8.8 mg/m^2 on an every 3-week cycle (21 days +/-2 days)
  All non-BSA based doses (flat dose) in Phase 2a were converted to BSA dosing units. Participants dosed under the initial MTD flat dosing regimen were assigned to the < 8.8 mg/m^2 or > 8.8 mg/m^2 dose groups based on the BSA conversion of the initial study flat dose.
Arm/Group | All Phase 2a Dose Expansion Participants
Number analyzed (Participants) | 66
mg/m^2 | 8.8

12. Secondary Outcome: Phase 2a: Progression Free Survival (PFS)
Description: Progression free survival (PFS) is defined as the time from the date of first dose of PEN-221 to the date of first documented disease progression per RECIST 1.1, or death due to any cause. If a participant had not progressed or died before the analysis cutoff date (31 Jul 2020), PFS was censored at the date of last adequate tumor assessment. Results based on Kaplan-Meier estimates.
Time Frame: From date of first treatment/trial entry until first documented progression or date of death from any cause, whichever came first, assessed up to data cutoff of 31 Jul 2020
Population: Outcome measured by cancer type. GI mid-gut NET, PNET, and SCLC participants enrolled into the study and who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2a Dose Expansion (GI Mid-gut NET Cohort) | Phase 2a Dose Expansion (PNET Cohort) | Phase 2a Dose Expansion (SCLC Cohort)
Number analyzed (Participants) | 32 | 15 | 19
Months | 9.0 [5.0 to 16.5] | 3.2 [2.0 to 5.9] | 1.4 [1.2 to 1.8]

13. Secondary Outcome: Phase 2a: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from the first dose of PEN-221 to the date of death due to any cause. If the participant had not died before data lock (31 Jul 2020), OS was censored at the date of last contact.
Time Frame: For each GI mid-gut NET, PNET, and SCLC, from date of first treatment/trial entry until the date of death from any cause, assessed up to data cutoff of 31 Jul 2020
Population: Outcome measured by cancer type. GI mid-gut NET, PNET, and SCLC patients enrolled into the study and who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2a Dose Expansion (GI Mid-gut NET Cohort) | Phase 2a Dose Expansion (PNET Cohort) | Phase 2a Dose Expansion (SCLC Cohort)
Number analyzed (Participants) | 32 | 15 | 19
Months | NA [13.1 to NA] — Median Overall Survival was not estimable at time of data lock (7 patients died and 25 were censored) | 21.0 [4.9 to 24.0] | 3.9 [1.8 to 5.5]

14. Secondary Outcome: Phase 2a: ORR for Gastrointestinal Mid-gut NETs (GI Mid-gut NET) and Pancreatic NETs (PNET)
Description: The Objective Response Rate (ORR) is defined as the proportion of patients with a best overall CR or PR as defined by RECIST 1.1 using the investigator assessment captured on the electronic Case Report Form.
Time Frame: For each GI mid-gut NET and PNET participant from the date of first treatment through the date of first documented progression, assessed up to data cutoff 31 Jul 2020
Population: Outcome measured by cancer type. GI mid-gut NET and PNET participants who received any amount of study drug and had at least 1 post-baseline efficacy assessment (RECIST 1.1).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2a Dose Expansion (GI Mid-gut NET Cohort) | Phase 2a Dose Expansion (PNET Cohort)
Number analyzed (Participants) | 26 | 12
Participants
  Responder | 0 | 0
  Non-Responder | 26 | 12

15. Secondary Outcome: Phase 2a: Duration of Response (DOR) for Gastrointestinal Mid-gut NETs (GI Mid-gut NET) and Pancreatic NETs (PNET)
Description: Duration of Response (DOR) is defined as the time from the first documented response (CR or PR), as assessed by the investigator, to the date of first documented disease progression or death due to underlying cancer. If a patient did not progress or die before the data cutoff date (31 Jul 2020), DOR was censored at the date of last adequate tumor assessment.
Time Frame: For each GI mid-gut NET and PNET participant, from the date of first treatment through the date of first documented progression, assessed up to data cutoff (31 Jul 2020)
Population: Outcome measured by cancer type. GI mid-gut NET cohort and PNET cohort participants who received any amount of study drug and had at least 1 post-baseline efficacy assessment (RECIST 1.1). No participants in the GI mid-gut NET cohort or PNET cohort had an objective response, so no data is presented for this Outcome Measure
Arm/Group | Phase 2a Dose Expansion (GI Mid-gut NET Cohort) | Phase 2a Dose Expansion (PNET Cohort
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Anti-PEN-221 Antibodies (ADA)
Description: Plasma Samples Using an Electrochemiluminescent Method for the Detection of Anti-PEN-221 Antibodies in Human Serum.
Time Frame: Baseline and every 6 weeks up to end of treatment for each patient.
Population: All participants who received any dose of study drug with at least 1 post-baseline immunogenicity assessment. Phase 2a participants dosed under the initial MTD dosing regimen were assigned to the < 8.8 mg/m^2 or > 8.8 mg/m^2 dose groups based on the BSA conversion of the initial study dose.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2a Dose Expansion (<8.8 mg/m^2): Participants in GINET, PNET, and SCLC received PEN-221 BSA calculated starting dose of less than8.8 mg/m^2 on an every 3-week cycle (21 days +/-2 days) All non-BSA based doses in Phase 2a were converted to BSA dosing units. Participants dosed under the initial MTD dosing regimen were assigned to the < 8.8 mg/m^2 or > 8.8 mg/m^2 dose groups based on the BSA conversion of the initial study dose.
Arm/Group | Phase 1 Dose Escalation (Cohort 1) | Phase 1 Dose Escalation (Cohort 2) | Phase 1 Dose Escalation (Cohort 3) | Phase 1 Dose Escalation (Cohort 4) | Phase 1 Dose Escalation (Cohort 5) | Phase 1 Dose Escalation (Cohort 6) | Phase 1 Dose Escalation (Cohort 7) | Phase 2a Dose Expansion (<8.8 mg/m^2) | Phase 2a Dose Expansion (8.8 mg/m^2) | Phase 2a Dose Expansion (>8.8 mg/m^2)
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 6 | 2 | 11 | 22 | 15
Participants
  Baseline ADA Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Baseline ADA Negative | 2 | 3 | 3 | 3 | 3 | 6 | 2 | 11 | 20 | 15
  ADA Positive On-Study Treatment | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 2
  Persistent Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Only Last Sample Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other Positive | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
  ADA Negative On-Study Treatment | 2 | 3 | 3 | 2 | 3 | 6 | 2 | 11 | 19 | 13

ADVERSE EVENTS:
Time Frame: From time of first dose of study drug through 28 days after the last dose of study drug for each participant up to data cut-off 31 Jul 2020.
Description: The Safety Analysis population was comprised of all enrolled patients who received any amount of study drug and have at least 1 post-baseline safety evaluation (AE, clinical laboratory assessments, vital signs, ECG (electrocardiogram), ECOG scores, physical examination). Participants were analyzed according to treatment received. Dose levels reported for Phase 2a Arms/Groups were collected for reporting in BSA format only.
Groups:
- Phase 1 Dose Escalation (Cohort 1): Participants in Cohort 1 received PEN-221 administered IV over 1 hour at the starting dose of 1.0 mg1 on an every 3-week cycle (21 days +/-2 days).
- Phase 1 Dose Escalation (Cohort 2): Participants in Cohort 2 received PEN-221 administered IV over 1 hour at the starting dose of 2.0 mg1 on an every 3-week cycle (21 days +/-2 days).
- Phase 1 Dose Escalation (Cohort 3): Participants in Cohort 3 received PEN-221 administered IV over 1 hour at the starting dose of 4.0 mg1 on an every 3-week cycle (21 days +/-2 days).
- Phase 1 Dose Escalation (Cohort 4): Participants in Cohort 4 received PEN-221 administered IV over 1 hour at the starting dose of 8.0 mg1 on an every 3-week cycle (21 days +/-2 days).
- Phase 1 Dose Escalation (Cohort 5): Participants in Cohort 5 received PEN-221 administered IV over 1 hour at the starting dose of 12.0 mg1 on an every 3-week cycle (21 days +/-2 days).
- Phase 1 Dose Escalation (Cohort 6): Participants in Cohort 6 received PEN-221 administered IV over 1 hour at the starting dose of 18.0 mg1 on an every 3-week cycle (21 days +/-2 days).
- Phase 1 Dose Escalation (Cohort 7): Participants in Cohort 7 received PEN-221 administered IV over 1 hour at the starting dose of 25.0 mg1 on an every 3-week cycle (21 days +/-2 days).
- Phase 2a Dose Expansion (<8.8 mg/m^2): Participants in GINET, PNET, and SCLC received PEN-221 BSA calculated starting dose of less than 8.8 mg/m^2 on an every 3-week cycle (21 days +/-2 days)
  All non-BSA based doses in Phase 2a were converted to BSA dosing units. Participants dosed under the initial MTD dosing regimen were assigned to the < 8.8 mg/m2 or > 8.8 mg/m2 dose groups based on the BSA conversion of the initial study dose.
- Phase 2a Dose Expansion (>8.8 mg/m^2): Participants in GINET, PNET, and SCLC received PEN-221 BSA calculated starting dose of more than 8.8 mg/m^2 on an every 3-week cycle (21 days +/-2 days)
  All non-BSA based doses in Phase 2a were converted to BSA dosing units. Participants dosed under the initial MTD dosing regimen were assigned to the < 8.8 mg/m2 or > 8.8 mg/m2 dose groups based on the BSA conversion of the initial study dose.
Arm/Group | Phase 1 Dose Escalation (Cohort 1) | Phase 1 Dose Escalation (Cohort 2) | Phase 1 Dose Escalation (Cohort 3) | Phase 1 Dose Escalation (Cohort 4) | Phase 1 Dose Escalation (Cohort 5) | Phase 1 Dose Escalation (Cohort 6) | Phase 1 Dose Escalation (Cohort 7) | Phase 2a Dose Expansion (<8.8 mg/m^2) | Phase 2a Dose Expansion (8.8 mg/m^2) | Phase 2a Dose Expansion (>8.8 mg/m^2)
All-Cause Mortality (participants affected / at risk) | 2/2 | 1/3 | 3/3 | 1/3 | 2/3 | 3/6 | 3/3 | 4/12 | 8/34 | 10/20
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/3 | 3/3 | 0/3 | 0/3 | 2/6 | 2/3 | 3/12 | 7/34 | 15/20
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 3/3 | 3/3 | 3/3 | 6/6 | 3/3 | 12/12 | 32/34 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Escalation (Cohort 1) (N=2) | Phase 1 Dose Escalation (Cohort 2) (N=3) | Phase 1 Dose Escalation (Cohort 3) (N=3) | Phase 1 Dose Escalation (Cohort 4) (N=3) | Phase 1 Dose Escalation (Cohort 5) (N=3) | Phase 1 Dose Escalation (Cohort 6) (N=6) | Phase 1 Dose Escalation (Cohort 7) (N=3) | Phase 2a Dose Expansion (<8.8 mg/m^2) (N=12) | Phase 2a Dose Expansion (8.8 mg/m^2) (N=34) | Phase 2a Dose Expansion (>8.8 mg/m^2) (N=20)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage intercranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic hemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Escalation (Cohort 1) (N=2) | Phase 1 Dose Escalation (Cohort 2) (N=3) | Phase 1 Dose Escalation (Cohort 3) (N=3) | Phase 1 Dose Escalation (Cohort 4) (N=3) | Phase 1 Dose Escalation (Cohort 5) (N=3) | Phase 1 Dose Escalation (Cohort 6) (N=6) | Phase 1 Dose Escalation (Cohort 7) (N=3) | Phase 2a Dose Expansion (<8.8 mg/m^2) (N=12) | Phase 2a Dose Expansion (8.8 mg/m^2) (N=34) | Phase 2a Dose Expansion (>8.8 mg/m^2) (N=20)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (9) | 1 (1) | 1 (2) | 2 (4) | 5 (10) | 2 (2) | 6 (7) | 16 (21) | 10 (17)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (7) | 1 (2) | 2 (2) | 2 (3) | 6 (15) | 0 (0) | 9 (15) | 15 (22) | 6 (10)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 13 (17) | 9 (13)
Abdominal Pain (Gastrointestinal disorders) | 1 (4) | 1 (8) | 1 (2) | 1 (2) | 0 (0) | 4 (13) | 1 (2) | 5 (8) | 7 (8) | 5 (9)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (3) | 2 (2) | 1 (3) | 1 (1) | 2 (4) | 2 (3) | 4 (8) | 8 (10) | 4 (10)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (9) | 1 (1) | 1 (4) | 2 (2) | 5 (11) | 0 (0) | 6 (9) | 16 (26) | 10 (17)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 3 (3) | 3 (5)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (4)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (2)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (4) | 0 (0) | 1 (5) | 1 (1) | 6 (7) | 11 (13) | 7 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 10 (15) | 6 (10)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 7 (8) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (13) | 0 (0) | 1 (1) | 5 (9) | 3 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (13) | 0 (0) | 1 (2) | 4 (5) | 2 (6)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (8) | 4 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (4) | 4 (6) | 1 (2) | 4 (12) | 10 (13) | 4 (5)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 8 (11) | 4 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 3 (4)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 3 (4) | 4 (6) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Hypoesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sixth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (3) | 3 (10) | 1 (1) | 3 (4) | 9 (12) | 9 (17)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (5) | 3 (9) | 1 (1) | 2 (3) | 7 (13) | 9 (17)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (5) | 10 (13) | 5 (8)
Blood creatinine increased (Investigations) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 7 (9) | 1 (2)
Weight decreased (Investigations) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 2 (3) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (10) | 3 (5)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 1 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (2)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalized ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pupil dilation procedure (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (6) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 6 (9) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 6 (10) | 3 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 7 (11) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 5 (6) | 5 (7)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 7 (10) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 2 (2) | 4 (4) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin tightness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 3 (12) | 0 (0) | 2 (2) | 7 (11) | 5 (12)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 7 (16) | 6 (11)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 2 (2) | 1 (3) | 1 (1) | 3 (4) | 6 (7)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may submit for publication or public disclosure based on the results of the study only after one of the following occurs as specified in the Clinical Trial Agreement:

1. Sponsor publication of the multi-center clinical trial results;
2. Sponsor notification that the multi-center clinical trial results submission is no longer planned; or
3. The eighteenth (18) month anniversary of the completion or early termination of the multi-center clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT02936323/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/23/NCT02936323/SAP_001.pdf